CLINICAL TRIAL: NCT03157596
Title: Effectiveness of an Oral Health Education Program for Caregivers of Children With Developmental Disabilities: A Cluster Randomized Trial
Brief Title: Oral Health Education for Caregivers of Children With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElTyeb, Sara Amir Hassan, M.D. (Individual)
Collaborators: Sudan Medical Specialization Board (SMSB) (Other Government); Elfatih Malik, MD (Unknown)
Responsible Party: Principal Investigator, Dr. Sara Amir Hassan ElTyeb, Dr. Sara Amir, ElTyeb, Sara Amir Hassan, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3600 - SMSB
Record Dates: First submitted 2017-05-13; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Developmental Disability
Keywords: disability; developmental disability; special healthcare needs
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): selected randomly from a list of all the 105 special education centers registered at the State Ministry of Education, and randomly allocated into intervention group.
  all the children with developmental disabilities in enrolled in the school who met the eligibility criteria were examined and all their parents were interviewed.
  Caregivers' baseline knowledge and attitudes towards the oral healthcare of their children was assessed by an interview questionnaire.
  examination for the children with developmental disabilities was carried out to assess caregivers' practice by assessing the oral hygiene level and amount of unmet treatment needs.
  educational intervention by an Oral Health Education Program for Caregivers of Children with developmental disabilities about the oral health care of Children with DD, in the form of a short video, accompanied by demonstration & followed by an interactive discussion .
  the same evaluation was carried out again 3 months after the intervention.
  Interventions: Other: Oral Health Educational Program for Caregivers of Children with developmental disabilities
- control group (No Intervention): Evaluation of the knowledge, attitude and practice of caregivers of children with developmental disabilities towards the oral health of their children at baseline and 3 months after without any intervention.

INTERVENTIONS:
Other: Oral Health Educational Program for Caregivers of Children with developmental disabilities — Oral Health Education Program for Caregivers of Children with developmental disabilities included information about health issues and obstacles encountered in children with DD & methods of prevention and management. It also emphasized on proper oral hygiene measures for this group. (University of Washington 2010)
  Arms: intervention group

SUMMARY:
Considering the impact of caregivers' oral health knowledge, attitudes and practices on the oral health of their children; we introduced an educational program to the parents and caregivers of children with developmental disabilities about the oral healthcare of their developmentally disabled children to rise up with the oral health status of those children.

DETAILED DESCRIPTION:
* Target Population; Parents of Children with DD enrolled in selected special education centers in Khartoum state, Khartoum, Sudan, and their developmentally disabled children.
* A convenient sample of two special education centers were selected randomly from a list of all the 105 special education centers registered at the State Ministry of Education, and allocated into intervention and control groups.
* One center was used as case who received the educational program and the other center was used as a control group.
* Eligibility Criteria: child aged 3-18, with a developmental disability, caregivers approval to participate (signed the informed consent).
* All the Children who met the eligibility criteria in both centers were examined and all their parents were interviewed, before and after the intervention.
* An interview questionnaire for the parents of Children with DD in both centers was used to evaluate their knowledge and attitude toward the oral health care of their children before and 3 months after the intervention.
* Oral examination was carried out to determine the baseline oral hygiene level and treatment needs of the Children with DD, before the educational session.
* A second examination was carried out after a period of 3 months after the educational session, to determine any change in oral hygiene and treatment needs of the children after their parents and or caregivers' attendance to the educational session.
* The baseline and follow up examination were carried out blindly by a calibrated dentist.
* The same examiner carried out the baseline and follow up examinations to avoid any inter-examiner variations.
* Oral examination was arranged according to oral health surveys basic methods recommended by WHO in 2013.
* The Simplified Oral Hygiene Index (measuring debris index and calculus index).
* Dentition Status and Treatment Needs chart provided in oral health assessment forms for children by the WHO 2013 was used to determine the amount of unmet dental needs and help in evaluating the caregivers' oral healthcare behaviours and the frequency of dental visits.

ELIGIBILITY:
Inclusion Criteria:

* has a developmental disability.
* enrolled in any of the randomly selected special education schools.
* caregivers signed the informed consent.

Exclusion Criteria:

* not a student in any of the randomly selected special education schools.
* caregivers refused to participate and sign the informed consent.
* age not in the range of 3 - 18 years old.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
improvement in oral hygiene status of children with developmental disabilities | 3 months
  simplified oral hygiene index recorded from the oral examination of children with disabilities are analyzed in cluster level for both intervention and control groups, and compared before and 3 months after the educational intervention.

SECONDARY OUTCOMES:
improvement in caregivers' knowledge about oral healthcare of their developmentally disabled children | 3 months
  score of knowledge recorded in the interview questionnaire to the caregivers of children with disabilities are analyzed in cluster level for both intervention and control groups, and compared before and 3 months after the educational intervention.
improvement in caregivers' attitude towards the oral healthcare of their developmentally disabled children | 3 months
  score of attitude recorded in the interview questionnaire to the caregivers of children with disabilities are analyzed in cluster level for both intervention and control groups, and compared before and 3 months after the educational intervention.
decrease in the unmet treatment needs of children with developmental disabilities | 3 months
  score of unmet treatment needs recorded from the oral examination of children with disabilities are analyzed in cluster level for both intervention and control groups, and compared before and 3 months after the educational intervention.

IPD SHARING:
Plan to Share IPD: Undecided